CLINICAL TRIAL: NCT02485847
Title: IRIS Registry: Intelligent Research in Sight Registry
Acronym: IRISRegistry
Status: Recruiting | Type: Observational
Sponsor: American Academy of Ophthalmology (Other)
Responsible Party: Sponsor
Other Study IDs: IRIS Registry
Record Dates: First submitted 2015-06-22; First posted 2015-06-30 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Eye Diseases
Keywords: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Ophthalmology — A registry of ophthalmic ambulatory encounters which captures essential data elements for continuous quality improvement efforts, enhanced patient care outcomes, and pay for performance programs.

SUMMARY:
The IRIS™ Registry (Intelligent Research in Sight) is the nation's first comprehensive eye disease clinical registry. The American Academy of Ophthalmology is developing it as part of the profession's shared goal of continual improvement in the delivery of eye care.The IRIS Registry will be a centralized system for ophthalmology practices to promote practice innovations and achieve clinical excellence.

DETAILED DESCRIPTION:
The IRIS Registry is primarily a clinical self-improvement tool. It will allow ophthalmologists to compare their patient outcomes, professional performance and care processes against other ophthalmologists across the country. The IRIS Registry will be able to measure the continuum of care from initial patient contact, through intervention and follow up.

Improve Patient Care - Monitor patient interactions, track interventions, identify and address gaps in quality of care, and measure quality outcomes.

Manage Patient Populations - Proactively manage clinical conditions for entire patient populations by running reports on specific care criteria.

Benchmark Your Practice - Identify practice strengths and weaknesses using the IRIS Registry's ophthalmology-specific clinical data from other practices to compare to the performance and outcomes data of your practice.

Run quality reports on demand - Providing clinician- and practice-level results, plus national results and patient-level detail for all IRIS Registry measures.

Enhance Quality and Practice Efficiency - Use the IRIS Registry data to analyze practice processes and procedures and as a source for fact-based decision-making. Because the IRIS Registry will capture data over time at the individual and practice level, it will help practices efficiently manage patient care and optimize practice resources.

Join a Community of Quality - Become a member of a like-minded community of quality-driven professionals striving to continuously improve patient care. Interact with your peers to create opportunities for sharing quality improvement strategies and broaden your professional network.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the denominator requirements for each measure.

Exclusion Criteria:

* None

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To ensure the IRIS Registry infrastructure is properly developed with features and functionalities that meets the needs of ophthalmologists, the IRIS Registry is currently only open to Academy members practicing in the United States and its territories.
Sampling Method: Non-Probability Sample
Enrollment: 20000000 (Estimated)
Dates: Start 2014-03; Primary Completion 2100-01 (Estimated); Study Completion 2100-01 (Estimated)

PRIMARY OUTCOMES:
Primary Open Angle Glaucoma (POAG): Optic Nerve Evaluation | Up to 5 years
  This measure is to be reported a minimum of once per reporting period for patients seen during the reporting period. It is anticipated that clinicians who provide the primary management of patients with primary open-angle glaucoma (in either one or both eyes) will submit this measure.
Age-Related Macular Degeneration (AMD): Dilated Macular Examination | Up to 5 years
  This measure is to be reported a minimum of once per reporting period for patients, aged 50 years and older, seen during the reporting period. It is anticipated that clinicians who provide the primary management of patients with age-related macular degeneration (in either one or both eyes) will submit this measure.
Diabetic Retinopathy: Documentation of Presence or Absence of Macular Edema and Level of Severity of Retinopathy | Up to 5 years
  Percentage of patients aged 18 years and older with a diagnosis of diabetic retinopathy who had a dilated macular or fundus exam performed which included documentation of the level of severity of retinopathy and the presence or absence of macular edema during one or more office visits within 12 months.
Diabetic Retinopathy: Communication with the Physician Managing On-going Diabetes Care | Up to 5 years
  Percentage of patients aged 18 years and older with a diagnosis of diabetic retinopathy who had a dilated macular or fundus exam performed with documented communication to the physician who manages the on-going care of the patient with diabetes mellitus regarding the findings of the macular or fundus exam at least once within 12 months.
Preventive Care and Screening: Influenza Immunization | Up to 5 years
  Percentage of patients, aged 6 months and older, seen for a visit between October 1 and March 31 who received an influenza immunization, or who reported previous receipt of an influenza immunization.
Pneumonia Vaccination Status for Older Adults | Up to 5 years
  Percentage of patients 65 years of age and older who have ever received a pneumococcal vaccine.
Diabetes Mellitus: Dilated Eye Exam in Diabetic Patient | Up to 5 years
  Percentage of patients aged 18 through 75 years with a diagnosis of diabetes mellitus who had a dilated eye exam.
Documentation of Current Medications in the Medical Record | Up to 5 years
  Percentage of patients aged 18 years and older with a list of current medications (includes prescription, over-the-counter, herbals, vitamin/mineral/dietary nutritional supplements) documented by the provider, including drug name, dosage, frequency and route
Melanoma: Continuity of Care - Recall System | Up to 5 years
  This measure is to be reported a minimum of once per reporting period for melanoma patients seen during the reporting period. It is anticipated that clinicians providing care for patients with melanoma or a history of melanoma will submit this measure.
Melanoma: Coordination of Care | Up to 5 years
  This measure is to be reported at each visit occurring during the reporting period for melanoma patients seen during the reporting period. It is anticipated that clinicians providing care for patients with melanoma will submit this measure.
Age-Related Macular Degeneration (AMD): Counseling on Antioxidant Supplement | Up to 5 years
  Percentage of patients aged 50 years and older with a diagnosis of AMD and/or their caregiver(s) who were counseled within 12 months on the benefits and/or risks of the Age-Related Eye Disease Study (AREDS) formulation for preventing progression of AMD
Primary Open-Angle Glaucoma (POAG): Reduction of Intraocular Pressure (IOP) by 15% or Documentation of a Plan of Care | Up to 5 years
  Percentages of patients aged 18 years and older with a diagnosis of POAG whose glaucoma treatment has not failed (the most recent IOP was reduced by at least 15% from the pre-intervention level) or if the most recent IOP was not reduced by at least 15% from the pre-intervention level, a plan of care was documented within 12 months.
Cataracts: 20/40 or Better Visual Acuity within 90 Days Following Cataract Surgery | Up to 5 years
  Percentage of patients aged 18 years and older with a diagnosis of uncomplicated cataract who had cataract surgery and no significant ocular conditions impacting the visual outcome of surgery and had best-corrected visual acuity of 20/40 or better (distance or near) achieved within 90 days following the cataract surgery.
Cataracts: Complications within 30 Days Following Cataract Surgery Requiring Additional Surgical Procedures | Up to 5 years
  Percentage of patients aged 18 years and older with a diagnosis of uncomplicated cataract who had cataract surgery and had any of a specified list of surgical procedures in the 30 days following cataract surgery which would indicate the occurrence of any of the following major complications; retained nuclear fragments, endophthalmitis, dislocated or wrong power intraocular lens, retinal detachment, or wound dehiscence.
Melanoma: Overutilization of Imaging Studies in Melanoma | Up to 5 years
  This measure is to be reported once per reporting period for patients with a current diagnosis of melanoma or a history of melanoma who are seen for an office visit during the reporting period. This measure is intended to reflect the quality of services provided for the primary management of patients with melanoma who have an office visit during the reporting period.
Preventive Care and Screening: Tobacco Use: Screening and Cessation Intervention | Up to 5 years
  Percentage of patients aged 18 years and older who were screened for tobacco use one or more times within 24 months and who received cessation counseling intervention if identified as a tobacco user.
Controlling High Blood Pressure | Up to 5 years
  Percentage of patients 18 through 85 years of age who had a diagnosis of hypertension and whose blood pressure was adequately controlled (< 140/90 mmHg) during the measurement period
Use of High-Risk Medications in the Elderly | Up to 5 years
  Percentage of patients aged 66 years and older who were ordered high-risk medications.
  Two rates are reported: 1. Percentage of patients who were ordered at least one high-risk medication. 2. Percentage of patients who were ordered at least two different high-risk medications.
Biopsy Follow-Up | Up to 5 years
  Percentage of patients whose biopsy results have been reviewed and communicated to the primary care/referring physician and patient by the performing physician
Improvement in Patient's Visual Function within 90 Days Following Cataract Surgery | Up to 5 years
  Percentage of patients aged 18 years and older in sample who had cataract surgery and had improvement in visual function achieved within 90 days following the cataract surgery, based on completing a pre-operative and postoperative visual function survey.
Patient Satisfaction within 90 Days Following Cataract Surgery | Up to 5 years
  Percentage of patients aged 18 years and older in sample who had cataract surgery and were satisfied with their care within 90 days following the cataract surgery, based on completion of the Consumer Assessment of Healthcare Providers and Systems Surgical Care Survey.
Falls: Screening for Future Fall Risk | Up to 5 years
  Percentage of patients 65 years of age and older who were screened for future fall risk during the measurement period.
Closing the Referral Loop: Receipt of Specialist Report | Up to 5 years
  Percentage of patients with referrals, regardless of age, for which the referring provider receives a report from the provider to whom the patient was referred.
Adult Primary Rhegmatogenous Retinal Detachment Repair Success Rate | Up to 5 years
  Percentage of surgeries for primary rhegmatogenous retinal detachment where the retina remains attached after only one surgery
Adult Primary Rhegmatogenous Retinal Detachment Surgery Success Rate | Up to 5 years
  Percentage of retinal detachment cases achieving flat retinas six months post surgery
Cataract Surgery with Intra-Operative Complications (Unplanned Rupture of Posterior Capsule requiring unplanned vitrectomy) | Up to 5 years
  Rupture of the posterior capsule during anterior segment surgery requiring vitrectomy
Cataract Surgery: Difference Between Planned and Final Refraction | Up to 5 years
  Percentage of patients who achieve planned refraction within +-1,0 D
Tobacco Use and Help with Quitting Among Adolescents | Up to 5 years
  The percentage of adolescents 12 to 20 years of age with a primary care visit during the measurement year for whom tobacco use status was documented and received help with quitting if identified as a tobacco user.
Corneal Graft: 20/40 or Better Visual Acuity within 90 Days following Corneal Graft Surgery | Up to 5 years
  Percentage of corneal graft surgery patients with a visual acuity of 20/40 or greater at 90 days after surgery
Open-Angle Glaucoma: Intraocular Pressure Reduction | Up to 5 years
  Percentage of glaucoma patient visits where their IOP was below a threshold level based on the severity of their diagnosis
Open-Angle Glaucoma: Visual Field Progression | Up to 5 years
  Percentage of eyes, in patients with a diagnosis of glaucoma, with a mean deviation loss of more than 3 decibels from their baseline value
Open-Angle Glaucoma: Intraocular Pressure Reduction Following Laser Trabeculoplasty | Up to 5 years
  Percentage of patients underwent laser trabeculoplasty who had IOP reduced by 20% from their pretreatment level
Acquired Involutional Ptosis: Improvement of Marginal Reflex Distance within 90 Days Following Surgery for Acquired Involutional Ptosis | Up to 5 years
  Percentage of surgical ptosis patients with an improvement of marginal reflex distance postoperatively
Acquired Involutional Entropion: Normalization of Eyelid Position within 90 Days Following Surgery for Acquired Involutional Entropion | Up to 5 years
  Percentage of surgical entropion patients with a postoperative normalized lid position
Amblyopia: Improvement of Corrected Interocular Visual Acuity Difference to 2 or fewer Lines | Up to 5 years
  Percentage of newly diagnosed amblyopic patients with a corrected interocular VA difference of 2 or fewer lines (< 0.23 logMAR) within 6 months of first diagnosis
Surgical Esotropia: Patients with Postoperative Alignment of 15 prism diopters or less | Up to 5 years
  Percentage of surgical esotropia patients with a postoperative alignment of 15 prism diopters or less
Diabetic Retinopathy: Dilated Eye Exam | Up to 5 years
  Percentage of patients aged 18 years and older with a diagnosis of diabetic retinopathy who had a dilated macular or fundus exam performed which included documentation of the level of severity of retinopathy and the presence or absence of macular edema during one or more office visits within 12 months
Exudative Age-Related Macular Degeneration: Loss of Visual Acuity | Up to 5 years
  Percentage of patients with a diagnosis of nonexudative age-related macular degeneration and taking AREDS supplements with of loss of less than 0.3 logMar of visual acuity within the past 12 months
Nonexudative Age-Related Macular Degeneration: Loss of Visual Acuity | Up to 5 years
  Percentage of patients with nonexudative age-related macular degeneration progressing to exudative age-related macular degeneration over the past 12 months
Diabetic Macular Edema: Loss of Visual Acuity | Up to 5 years
  Percentage of patients with a diagnosis of diabetic macular edema with of loss of less than 0.3 logMar of visual acuity within the past 12 months
Rhegmatogenous Retinal Detachment Surgery: Visual acuity improvement within 90 days of surgery | Up to 5 years
  Percentage of patients who underwent rhegmatogenous retinal detachment surgery and achieved an improvement in their visual acuity from their preoperative level within 90 days of surgery in the treated eye.
Rhegmatogenous Retinal Detachment Surgery: Return to the operating room within 90 days of surgery | Up to 5 years
  Percentage of patients who underwent rhegmatogenous retinal detachment surgery and had a return to the operating room within 90 days
Acute Anterior Uveitis: Post-treatment visual acuity | Up to 5 years
  Percentage of acute anterior uveitis patients with a post-treatment best corrected visual acuity of 20/40 or greater OR patients whose visual acuity had returned to their baseline value prior to onset of uveitis
Acute Anterior Uveitis: Post-treatment Grade 0 anterior chamber cells | Up to 5 years
  Percentage of patients with acute anterior uveitis post-treatment with Grade 0 anterior chamber cells
Chronic Anterior Uveitis: Post-treatment visual acuity | Up to 5 years
  Percentage of chronic anterior uveitis patients with a post-treatment best corrected visual acuity of 20/40 or greater OR patients whose visual acuity had returned to their baseline value prior to onset of uveitis
Chronic Anterior Uveitis: Post-treatment Grade 0 anterior chamber cells | Up to 5 years
  Percentage of patients with chronic anterior uveitis post-treatment with Grade 0 anterior chamber cells

CONTACTS AND LOCATIONS:
Overall Officials: Flora Lum, MD, Study Director — American Academy of Ophthalmology
Locations (1):
- American Academy of Opthalmology, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IRIS Registry web site — http://www.aao.org/irisregistry